CLINICAL TRIAL: NCT02154295
Title: Simultaneous Acquisition of Intravascular Ultrasound and Near Infrared Spectroscopy Data in the Coronary Artery Study
Brief Title: In Vitro and In Vivo Comparison Between Intravascular Ultrasound (IVUS) Systems
Acronym: SAVOIR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Infraredx (Industry)
Collaborators: South Australian Health and Medical Research Institute (Other); Royal Adelaide Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 0126
Record Dates: First submitted 2014-05-16; First posted 2014-06-03 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eagle Eye Platinum (Active Comparator): Eagle Eye Platinum Catheter as the comparator.
  Interventions: Device: Infraredx Test Catheter
- Revolution (Active Comparator): Revolution Catheter as the comparator
  Interventions: Device: Infraredx Test Catheter
- TVC Insight 40MHz (Active Comparator): TVC Insight as comparative catheter.
  Interventions: Device: Infraredx Test Catheter
- Atlantis Pro (Active Comparator): Atlantis Pro catheter as comparator
  Interventions: Device: Infraredx Test Catheter

INTERVENTIONS:
Device: Infraredx Test Catheter

SUMMARY:
The purpose of this study is to investigate and compare the images obtained from coronary imaging catheters used in the treatment of coronary blockages both in a clinical setting with patients and in models.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Scheduled for a coronary angiogram at the Royal Adelaide Hospital.
* Women must be non-lactating or not of childbearing potential (1 year post menopausal or surgically sterilized [total hysterectomy, bilateral tubal ligation, bilateral oophorectomy]).
* Target artery must be >2 mm to accommodate the IVUS catheter.
* IVUS must be clinically indicated or indeterminate angiographic lesion in the artery (40%-70% angiographic stenosis)

Exclusion Criteria:

* Cardiogenic shock
* Contraindications to intracoronary nitroglycerin (hypertrophic obstructive cardiomyopathy; cerebral hemorrhage, head trauma; concomitant sildenafil, tadalafil or vardenafil use)
* Known coronary artery spasm
* Significant bleeding risk (i.e. previous hemorrhagic stroke, active peptic ulcer disease)
* Bleeding diathesis
* Significant renal impairment (patients will be excluded if their calculated creatinine clearance is < 30 mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Clarity of Image and ease of interpretation as measured by physician survey | Day 0

SECONDARY OUTCOMES:
Comparison of diameters and areas using ultrasound imaging from a standard test fixture(model) and test catheters | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sidharta, MBBS BMedSc, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia